CLINICAL TRIAL: NCT01978795
Title: The Effectiveness of a Web-Based Resource in Improving Post-Concussion Management in High Schools
Brief Title: Interactive Training in Sports Concussion Prevention and Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ann Glang, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HD056610; R44HD056610 (NIH)
Record Dates: First submitted 2013-10-23; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-10

CONDITIONS: Concussion
Keywords: concussion; high school; web-based training; school-based health care
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brain 101 website (Experimental): Brain 101: The Concussion Play book is a web-based, stand-alone guide for school leaders on effective policies and practices in concussion management. The website offers a school-wide approach to preventing and managing sports concussion, including a) training for educators, athletics staff, students, and parents; b) guidelines for creating a concussion management team; and c) information on strategies for supporting students in the classroom following concussion.
  Interventions: Other: Brain 101 website
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Brain 101 website — Brain 101: The Concussion Play book is a web-based, stand-alone guide for school leaders on effective policies and practices in concussion management. Consistent with the literature on effective school-based change efforts, the website offers a comprehensive, school-wide approach to preventing and managing sports concussion, including training for educators, athletics staff, students, and parents. The website presents guidelines for creating a concussion management team (CMT) that meets regularly to support students as they return to academics, extra-curricular activities, and athletics. It also includes information on strategies for supporting students in the classroom following concussion (e.g., designing reduced school schedules, monitoring school performance following concussion).
  Arms: Brain 101 website
Other: Control — At control schools, parents viewed Centers for Disease Control materials on safe teen drivers. Athletes viewed web-based materials about teens staying safe on the job.
  Arms: Control

SUMMARY:
This study evaluated Brain 101: The Concussion Play book, an intervention that provides education and resources on concussion management for high schools. The study hypotheses were that athletes and parents who viewed the Brain 101 program would demonstrate increased knowledge and self efficacy in concussion management, and that use of the intervention would positively affect school concussion management practices.

ELIGIBILITY:
Inclusion Criteria for participating schools:

* athletic trainer (AT) on staff or contracted by school for services
* school access to a high-speed internet connection
* agreement to expose all students participating in fall sports to the training.

Exclusion Criteria:

* didn't meet inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change in youth athlete and parent knowledge of effective sports concussion management from before and after intervention exposure | Pre: Participants completed the measure an average of 30 minutes prior to being exposed to the intervention. Post: Participants completed the measure an average of 30 minutes after exposure to the intervention

SECONDARY OUTCOMES:
Change in youth athlete and parent ratings of self-efficacy in sports concussion management | Pre: Participants completed the measure an average of 30 minutes prior to being exposed to the intervention. Post: Participants completed the measure an average of 30 minutes after exposure to the intervention

OTHER OUTCOMES:
Implementation of effective concussion management guidelines | 3 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ann E Glang, PhD, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States

REFERENCES:
- [Derived] Glang AE, Koester MC, Chesnutt JC, Gioia GA, McAvoy K, Marshall S, Gau JM. The effectiveness of a web-based resource in improving postconcussion management in high schools. J Adolesc Health. 2015 Jan;56(1):91-7. doi: 10.1016/j.jadohealth.2014.08.011. Epub 2014 Oct 29. PMID 25438964